CLINICAL TRIAL: NCT03824925
Title: Efficacy of Zinc Sulfate on Concurrent Chemoradiotherapy Induced Taste Alterations in Oral Cancer Patients- A Double Blind Randomized Controlled Trial
Brief Title: Efficacy of Zinc on Concurrent Chemo-radiotherapy Induced Taste Alterations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Asma Hayat Khan, Post Graduate Trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHKhan
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Taste, Altered
Keywords: Taste alterations; zinc sulfate; oral cancer; taste acuity
MeSH Terms: conditions — Dysgeusia; Mouth Neoplasms | interventions — Starch; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each patient was asked to pick one of the sealed envelopes from a box. The sealed envelopes contained either alphabets A or B. The sealed envelopes were blinded to both the investigator and the patient. The generation of random allocation sequence and assignment of participants to intervention were done by the principal investigator.
  Both the investigator and the patient were blinded (double-blinded) about the groups and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo oral zinc capsules (Placebo Comparator): Group A: It was the control group. Participants were advised to start taking placebo capsule of Zinc in a look alike preparation on their first day of chemo-radiotherapy and continued taking it a month after their chemo-radiotherapy ended
  Interventions: Drug: Placebo oral Zinc capsule; Drug: Zinc Sulfate 220 MG
- Zinc Sulfate 220 MG (Experimental): Group B: Cap zinc 220 mg (equivalent to 50 mg of elemental zinc) on 1st day of their chemo-radiotherapy and continued taking it a month after their chemo-radiotherapy ended.
  Interventions: Drug: Placebo oral Zinc capsule; Drug: Zinc Sulfate 220 MG

INTERVENTIONS:
Drug: Placebo oral Zinc capsule — Look alike cap of corn starch as a placebo of Zinc to be given on day 1 of chemo-radiotherapy
  Other Names: Corn Starch
Drug: Zinc Sulfate 220 MG — Zinc sulfate in test group dose was 220 mg which is equivalent to 50 mg of elemental zinc
  Other Names: Zincat

SUMMARY:
Taste changes are common in cancer patients receiving concurrent chemoradiation which become a significant complaint and a cause of distress and morbidity. Loss of gustatory function further advances to malnutrition, weight loss, reduced quality of life, poor compliance and even diminished response to drug therapy. Taste is an essential sensation which serves oral intake of food and enables to prevent the ingestion of potentially harmful and poisonous substances. The sense of taste is crucial for an individual's well-being and psychological health. Taste changes may advance to reduced appetite, dietary insufficiency, food repulsion affecting body weight and anorexia further leading to impaired immunity, decline in health status and malnutrition. As taste impairment is not a life-threatening event therefore it might not be reported by some patients. Hence, this aspect is neglected despite being a common and distressing side-effect of chemoradiation. Due to the location of the cancer and the long-term effects of cancer therapies, patients with oral cavity cancers have a specially high prevalence of chemosensory disorders. Zinc is comparatively non-toxic if taken orally, and rather non-toxic in contrast to other trace metals such as manganese and iron. Zinc is an integral element in both the maintenance and repair of taste buds. It is involved in promoting the diffusion of taste stimuli to taste buds. Salivary zinc has been found in association with Gustin (carbonic anhydrase, CA VI), a zinc-metalloprotein enzyme that may be involved with providing nutrition to the human taste buds. Zinc influences the synthesis of gustin required for the growth, development, maintenance and production of taste buds and regulation of taste function.

The hypothesis was:

Null hypotheses: There is no difference in the taste acuity between test and control group with the administration of zinc sulfate.

Alternative hypotheses: There is a difference in the taste acuity between test and control group with the administration of zinc sulfate.

Thus, the present study aimed to observe changes in taste function of oral cancer patients by detection and recognition thresholds before beginning their treatment (before chemoradiation and intervention), at the end of chemoradiation and a month after and to evaluate the preventive effect of zinc sulfate on chemoradiation-induced taste changes. To the best of our knowledge, similar study has not been conducted before in our region.

DETAILED DESCRIPTION:
Consecutive Sampling was used. It was a two-stage sampling method. Data was collected from patients visiting the Oncology Section at Atomic Energy Medical Centre Karachi from September 2017 to March 2018 on a proforma after being examined by the section head oncologist for the tumor. A standard proforma was used to record the taste acuity of the participants. Furthermore, the proforma also had details about patient's site of tumor, stage of tumor, daily fraction of dose, total dose of radiotherapy, chemotherapeutic drug and duration of the treatment for the record.

The international Standard Organization ISO 3972:2011/Cor 1:2012 provides guidelines for Method of investigating sensitivity of taste. Therefore, all solutions were prepared in accordance with the ISO. The solutions were prepared with deionized water in grams/litre and stored in 1000ml glass bottles at room temperature. All solutions were colorless and odorless. Eight increasing concentration of each taste (salty, sweet, sour and bitter; altogether 32 bottles), zinc capsules and placebo (filled with cornstarch) were prepared by ATCO pharmaceuticals. Sodium chloride was used as a stimulus for salty, sucrose for sweet, citric acid for sour and caffeine for bitter.

Patients were instructed to refrain from eating or drinking 30 mins to 1 hour before the procedure. If any patient was wearing denture it was taken off before the procedure and mouth was thoroughly rinsed with water before each trial. Each subject was given single 15ml of each solution in a cup and asked to hold the solution for 30 seconds in their mouth and gargle out to make sure the whole of oral cavity will be exposed to the taste solution (sip and spit procedure). After each presentation, patient mouth was thoroughly rinsed with water to remove any after taste and to avoid the residual effect of the previous taste solution. The water used for rinsing was identical with that used for preparing solutions. Each trial was spaced at least 15 seconds apart. The time spent for each data collection tool was 20-30 mins.

Taste function of each patient for four basic taste (salty, sweet, sour and bitter) was assessed by detection and recognition threshold which were noted on a proforma. The proforma had three columns (baseline, end chemoradiation and follow-up a month after chemoradiation) for each taste and marking from 1 to 8 corresponding to the increasing concentration of the taste solutions (D8-D1) for each taste. D1 was considered as the highest concentration whereas D8 was the lowest concentration of each taste solution.

The cut-off values that were set for each patient for detection and recognition threshold were:

1-8 = able to identify and recognize the taste 0 = unable to identify and recognize any response For Detection threshold (DT) A sample of deionized water and a taste sample was presented to the patient. The order of presentation was randomized for every subject. Participants were asked to indicate which of the sample contains the taste. Detection threshold (DT) was considered as the lowest level at which a subject can perceive a stimulus. This was the minimum concentration at which the subject can detect that there is something different from water, but may not identify its quality. D1 was the highest concentration of solution for each taste and was marked on proforma as 1 and D8 was the minimum concentration and was marked as 8.

For Recognition threshold (RT) Participants were also asked to describe the taste of the solution either salty, sweet, sour or bitter. Recognition threshold was considered as the lowest level of a solution at which a subject can correctly recognize its taste, i.e., sucrose for sweet, sodium chloride (NaCl) for salty, citric acid for sour and caffeine for bitter. D1 was the highest concentration of solution for each taste and was marked as 1 whereas D8 was the minimum concentration and was marked as 8.

Solutions were presented in the increasing order of their concentration and the lowest concentration of solution was marked for each taste that was perceived by the patient. Any subject who was unable to detect the difference between the water and the tastant, the concentration of the taste solution was increased.

Data was entered and analyzed by the IBM SPSS software for windows version 20. Data is shown as mean ± SD for descriptive statistics and as median [IQR] for intervention statistics. First, the normality was assessed of all four taste variables by Shapiro-Wilk test. The normality tests are given below.

The baseline characteristics of the test and control group were compared by Chi square and independent t test. To observe difference within the two groups, Wilcoxon Signed Ranks test was applied. To observe the difference between the two groups, Mann-Whitney U test was used. P-value was calculated by Friedman test. Statistical significance was accepted at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Oral cancer patients undergoing concurrent chemotherapy with radiotherapy for the first time as a single treatment modality.
* Patients aged between 20-60 years.
* Radiation planned between 60-70 Gy of external beam radiotherapy.
* Cisplatin as primary chemotherapeutic agent.

Exclusion Criteria:

* Previous history of radiotherapy or chemotherapy regardless of time.
* Existence of oral lesions such as aphthous ulcers, stomatitis or candidosis at the time of selection.
* Cranial nerve lesions of V, VII, IX and partial or total glossectomy.
* Individuals with nose or ear infections which can influence taste, metabolic or endocrine disorders that may affect taste sensitivity (Sjogren syndrome, hypertension, diabetes mellitus, renal disease, liver disease and thyroid disease).
* Concomitant administration of a drug with Chemoradiation which may affect taste (metronidazole, diuretics and anti-depressants).
* Individuals already on medications associated with taste disturbances such as penicillamine, tetracyclines, quinolones, and bisphosphonates for any existing condition.
* Patients who didn't agree to participate and sign consent form and lack of cooperation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Change in taste acuity with the administration of zinc sulfate in oral cancer patients receiving chemo-radiotherapy by detection and recognition threshold on a proforma | Taste acuity was observed for each taste at 3 stages that is, Baseline: before starting chemo-radiotherapy, after 7-8 week (on last day of chemo-radiotherapy), 11-12 week (follow-up after 1 month of their therapy)
  Every participant's taste acuity was by detection and recognition using different concentrations of taste solutions. The solutions were prepared in accordance with the International Standard Organization 3972:2011/Cor 1:2012 which provides guidelines for Method of investigating of taste sensitivity. Sodium chloride was used as a stimulus for salty, sucrose for sweet, citric acid for sour and caffeine for bitter. Detection threshold was the minimum concentration at which the subject can detect that there is something different from water, but may not identify its quality. Recognition threshold was considered as the lowest level of a solution at which a subject can correctly recognize its taste.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Khan, MSc-DS, Principal Investigator — Dow Ishrat ul Ebad Institute of Oral Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided